CLINICAL TRIAL: NCT06874504
Title: Clinical Validation of the Norbert Health Device for Pulse Rate Measurement
Status: Completed | Type: Observational
Sponsor: Norbert Health (Industry)
Collaborators: Integrative Clinical Trials, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: NCP-0004
Record Dates: First submitted 2025-03-06; First posted 2025-03-13 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Norbert Device — The Norbert Device (ND) is a contactless, noninvasive device that provides measurements of pulse rate.

SUMMARY:
The study will evaluate the measuring pulse rate (PR) using the Norbert Device (ND) as compared to a reference heart rate measured using an electrocardiogram (ECG).

DETAILED DESCRIPTION:
The study design is to validate the pulse rate accuracy. The study is a non-randomized, non-blinded single arm design to evaluate the clinical accuracy of the ND's pulse rate measurement compared to a reference heart rate manually measured by observing R-peaks in a standard concurrently recorded ECG from an FDA 510(k)-cleared reference clinical ECG (RCECG). The sponsor will ensure that the study staff enrolls a range of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years or older
* Ability to comprehend written consent and provide informed consent
* Ability to commit to and complete study related paperwork and activities (i.e. subject forms, have de-identified pictures taken, comply with periods of no movement, etc.)

Exclusion Criteria:

* Pregnant women
* Diagnosis of essential tremor or any medical condition causing tremors of the head or hands
* Facial tattoos, scars, large moles, beards/hair growth, birthmarks, vitiligo, skin conditions, facial discoloration, or heavy makeup within the areas of interest
* Inability for subject to avoid extreme movement during measurement reading windows
* Inability for subject to raise their hand during measurement reading windows
* No heart arrythmias
* Discretion of the Principal investigator or clinical study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects 18 years of age or older with the ability to consent to study and follow instructions needed for data collection. Data will be collected on enrolled patients including but not limited to diabetes, hypertension, cardiac conditions, circulation problems, medications, and other health issues that would affect blood circulation to skin. Subject enrollment for these comorbidities and others will be based on incidental enrollment from the pool of available subjects per site.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Primary Objective | Approximately 1 hour
  To validate the accuracy specification for pulse rate from the ND when compared to an FDA-cleared medical device for heart rate monitoring electrocardiogram (ECG monitor, 5 lead).

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Clinical Trials, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No